CLINICAL TRIAL: NCT02907918
Title: A Phase II Neoadjuvant Study of Palbociclib in Combination With Letrozole and Trastuzumab as Neoadjuvant Treatment of Stage II-III ER+ HER2+ Breast Cancer (PALTAN)
Brief Title: Neoadjuvant Study of Palbociclib in Combination With Letrozole and Trastuzumab in Stage II-III ER+ HER2+ Breast Cancer
Acronym: PALTAN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility
Sponsor: Washington University School of Medicine (Other)
Collaborators: Pfizer (Industry); Rising Tide Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201610019
Record Dates: First submitted 2016-09-14; First posted 2016-09-20 (Estimated); Results first posted 2021-09-05 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer; Cancer of Breast; Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Letrozole; Trastuzumab; Goserelin; Mastectomy, Segmental; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Palbociclib + letrozole + trastuzumab +/- goserelin (Experimental): * Neoadjuvant palbociclib + letrozole (plus goserelin if premenopausal) + trastuzumab for a total of 16 weeks, consisting of (4) 28-day cycles
  * Definitive surgery will be performed preferably within 6 weeks after the end of Cycle 4. Letrozole and trastuzumab will continue until the day of surgery. Letrozole will continue to be taken daily and trastuzumab will be given every 3 weeks per standard of care guidelines. Adjuvant therapy following definitive surgery will be at the discretion of the treating physician
  Interventions: Drug: Palbociclib; Drug: Letrozole; Biological: Trastuzumab; Drug: Goserelin; Procedure: Breast surgery; Procedure: Research tumor biopsy; Procedure: Research bone marrow (OPTIONAL); Procedure: Research blood sample; Genetic: Research blood for germline DNA; Procedure: Blood for detection of circulating tumor cells

INTERVENTIONS:
Drug: Palbociclib — Palbociclib is an oral drug given at a dose of 125 mg daily on Days 1-21 of each 28-day cycle for a total of 4 cycles.
  Other Names: Ibrance
Drug: Letrozole — Letrozole is an oral drug given at a dose of 2.5 mg orally once a day. It will be taken continuously (Days 1-28 of each cycle) until the day of definitive surgery.
  Other Names: Femara®
Biological: Trastuzumab — * Or FDA approved biosimilar
  * Trastuzumab will be administered on a weekly basis for 16 weeks (on Days 1, 8, 15, and 22 of each 28-day cycle for a total of 4 cycles). The first dose of trastuzumab on Cycle 1 Day 1 will be a loading dose of 4 mg/kg IVPB over 90 minutes. Subsequent doses of trastuzumab will be 2 mg/kg IVPB over 30 minutes. Weekly trastuzumab will continue after the completion of Cycle 4 of palbociclib until surgery.
  Other Names: Herceptin®
Drug: Goserelin — Goserelin is given subcutaneously at a dose of 3.6 mg on Day 1 of each cycle. Goserelin will be continued (once every 28-days) after the completion of Cycle 4 of palbociclib if required.
  Other Names: Zoladex
Procedure: Breast surgery — Standard of care
Procedure: Research tumor biopsy — Baseline, cycle 1 day 15, and surgery
Procedure: Research bone marrow (OPTIONAL) — Baseline and surgery
Procedure: Research blood sample — Baseline, cycle 1 day 15, surgery, and yearly post-surgery for 5 years
Genetic: Research blood for germline DNA — Baseline
Procedure: Blood for detection of circulating tumor cells — Baseline

SUMMARY:
The investigators propose to influence estrogen receptor (ER) signaling by combining endocrine therapy with CDK4/6 inhibition along with trastuzumab in ER+/ human epidermal growth factor receptor 2 (HER2)+ early stage breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed clinical stage II or III ER+/HER2+ breast cancer with complete surgical excision of the breast cancer after neoadjuvant therapy as the treatment goal, staging criteria is to be based on AJCC 7.
* Tumor size at least 2 cm in one dimension by clinical or radiographic exam (World Health Organization (WHO) criteria). Patients with histologically confirmed palpable lymph nodes may be enrolled regardless of breast tumor size. A palpable mass is not required as long as the mass is at least 2 cm in one dimension by radiographic exam.
* At least 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* Normal bone marrow and organ function as defined below:

  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcl
  * Platelets ≥ 100,000/mcl
  * Total bilirubin ≤ institutional upper limit of normal (IULN)
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN
* Creatinine ≤ IULN OR creatinine clearance ≥ 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Left ventricular ejection fraction (LVEF) ≥ 50% by transthoracic echocardiogram or multigated acquisition scan (MUGA)
* Baseline corrected QT interval (QTcF) < 480 ms
* Women of childbearing potential must agree to undergo pregnancy testing within 14 days of study entry and agree to use adequate contraception (barrier method of birth control, abstinence, not hormonal) prior to study entry and for the duration of study participation as well as chemical LHRH Agonist with goserelin. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Prior systemic therapy for indexed breast cancer.
* Indeterminate or negative HER2 status.
* Inflammatory breast cancer.
* A history of other malignancy ≤ 5 years from diagnosis of indexed BC with the exception of basal cell or squamous cell carcinoma of the skin treated with local resection only or carcinoma in situ of the cervix.
* Currently receiving any other investigational agents or received any within the past 28 days.
* Know to be HIV positive.
* Known hepatitis B or C infection.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to palbociclib, letrozole, trastuzumab, any other aromatase inhibitor, any other monoclonal antibody, or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Current use or anticipated need for food or drugs that are known strong CYP3A4 inhibitors (i.e., grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, posaconazole, erythromycin, clarithromycin, telithromycin, indinavir, saquinavir, ritonavir, nelfinavir, lopinavir, atazanavir, amprenavir, fosamprenavir, nefazodone, diltiazem, and delavirdine) or inducers (i.e. dexamethasone, glucocorticoids, progesterone, rifampin, phenobarbital, St. John's wort).
* Any condition that impairs the ability to swallow or absorb oral medication (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affective absorption).
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2020-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Foluso O Ademuyiwa, M.D, MPH, Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - Mayo Clinic, Phoenix, Arizona
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ademuyiwa FO, Northfelt DW, O'Connor T, Levine E, Luo J, Tao Y, Hoog J, Laury ML, Summa T, Hammerschmidt T, Guo Z, Frith A, Weilbaecher K, Opyrchal M, Aft R, Clifton K, Suresh R, Bagegni N, Hagemann IS, Iglesia MD, Ma CX. A phase II study of palbociclib plus letrozole plus trastuzumab as neoadjuvant treatment for clinical stages II and III ER+ HER2+ breast cancer (PALTAN). NPJ Breast Cancer. 2023 Jan 6;9(1):1. doi: 10.1038/s41523-022-00504-z. PMID 36609389
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Palbociclib + Letrozole + Trastuzumab +/- Goserelin
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Palbociclib + Letrozole + Trastuzumab +/- Goserelin
Number analyzed (Participants) | 26
Age, Continuous [Median (Full Range); unit: years] | 59 [32 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pathologic Complete Response (pCR)
Description: A pathologic complete response (pCR) is defined as no histology evidence of invasive tumor cells in the surgical breast specimen and sentinel or axillary lymph nodes.
Time Frame: Completion of 4 cycles of treatment (approximately 16 weeks)
Population: One participant is not evaluable for this outcome measure because the participant experienced progressive disease after completion of treatment but prior to surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Letrozole + Trastuzumab +/- Goserelin
Number analyzed (Participants) | 25
Participants | 2

2. Secondary Outcome: Safety and Tolerability of Palbociclib in Combination With Neoadjuvant Letrozole and Trastuzumab (or FDA Approved Biosimilar) as Measured by Number of Participants With Grade 3 & 4 Adverse Events
Description: -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
Time Frame: 30 days after completion of neoadjuvant therapy (approximately 21 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Letrozole + Trastuzumab +/- Goserelin
Number analyzed (Participants) | 26
Participants
  Neutrophil count decreased | 13
  Lymphocyte count decreased | 1
  Hypertension | 8
  White blood cell decreased | 2
  Colitis | 1
  Hypokalemia | 1
  Pulmonary edema | 1
  Ventricular tachycardia | 1
  Alanine aminotransferase increased | 1
  Aspartate aminotransferase increased | 1
  Colonic obstruction | 1

3. Secondary Outcome: Change in Patient Reported Outcomes as Measured by NCI PRO-CTCAE
Description: * Answers ranging from None to Very Severe (none=0 to very severe=4); Not at All to Very Much (not at all=0 to very much=4), Never to Almost Constantly (0=never to almost constantly=4)
  * PRO-CTCAE responses are scored from 0 to 4, and there are no standardized scoring rules yet established for how to combine attributes into a single score or how best to analyze PRO-CTCAE data longitudinally.
  * PRO-CTCAE scores for each attribute (frequency, severity and/or interference) will be presented descriptively
Time Frame: Baseline, cycle 2 day 1 (approximately 29 days), and end of cycle 4 (approximately 16 weeks)
Population: 3 participants at the end of cycle 4 did not complete the questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline: Palbociclib + Letrozole + Trastuzumab +/- Goserelin; Cycle 2 Day 1: Palbociclib + Letrozole + Trastuzumab +/- Goserelin; End of Cycle 4: Palbociclib + Letrozole + Trastuzumab +/- Goserelin: * Neoadjuvant palbociclib + letrozole (plus goserelin if premenopausal) + trastuzumab for a total of 16 weeks, consisting of (4) 28-day cycles
  * Definitive surgery will be performed preferably within 6 weeks after the end of Cycle 4. Letrozole and trastuzumab will continue until the day of surgery. Letrozole will continue to be taken daily and trastuzumab will be given every 3 weeks per standard of care guidelines. Adjuvant therapy following definitive surgery will be at the discretion of the treating physician
Arm/Group | Baseline: Palbociclib + Letrozole + Trastuzumab +/- Goserelin | Cycle 2 Day 1: Palbociclib + Letrozole + Trastuzumab +/- Goserelin | End of Cycle 4: Palbociclib + Letrozole + Trastuzumab +/- Goserelin
Number analyzed (Participants) | 26 | 26 | 23
score on a scale
  In the last 7 days, what was the severity of your decreased appetite at its worst? | 1.3461538 (0.8918434) | 1.3461538 (0.6894814) | 1.3043478 (0.8756703)
  In the last 7 days, how much did decreased appetite interfere with your usual or daily activities? | 1.0769231 (0.8448942) | 0.9615385 (0.3441824) | 1.0434783 (0.3665888)
  In the last 7 days, how often did you have nausea? | 1.2307692 (0.5870395) | 1.5000000 (0.9899495) | 1.2608696 (0.5408236)
  In the last 7 days, what was the severity of your nausea at its worst? | 1.1923077 (0.800961) | 1.4230769 (0.8566482) | 1.2173913 (0.6712622)
  In the last 7 days, what was the severity of your shortness of breath (SOB) at its worst? | 1.1923077 (0.5670436) | 1.1153846 (0.515901) | 1.4347826 (0.8957519)
  In the last 7 days, how much did your SOB interfere with your usual or daily activities? | 0.9615385 (0.4454902) | 1.0384615 (0.4454902) | 1.173913 (0.6503268)
  In the last 7 days, what was the severity of your cough at its worst? | 1.1923077 (0.4019185) | 1.2307692 (0.5870395) | 1.5217391 (1.0816471)
  In the last 7 days, how much did your cough interfere with your usual and daily activities? | 1.0000000 (0.2828427) | 1.0384615 (0.5276946) | 1.3043478 (0.9739695)
  In the last 7 days, how often did you have arm or leg swelling? | 1.0000000 (0.0000000) | 1.0384615 (0.3441824) | 1.2608696 (0.9153832)
  In the last 7 days, what was the severity of your arm or leg swelling at its worst? | 0.8846154 (0.3258126) | 1.0384615 (0.5276946) | 1.1304348 (0.4576966)
  In the last 7 days, how much did arm or leg swelling interfere with your usual or daily activities? | 0.9230769 (0.2717465) | 0.8846154 (0.3258126) | 1.0434783 (0.474654)
  In the last 7 days, how often did you feel a pounding or racing heartbeat (palpitations)? | 1.1538462 (0.4640955) | 1.1923077 (0.5670436) | 1.173913 (0.4910262)
  In the last 7 days, what was the severity of your pounding or racing heartbeat at its worst? | 1.0384615 (0.4454902) | 1.1923077 (0.6939297) | 1.1304348 (0.5480833)
  In the last 7 days, did you have any rash? | 1.8461538 (0.3679465) | 1.6153846 (0.5710988) | 1.826087 (0.3875534)
  In the last 7 days, what was the severity of your dry skin at its worst? | 1.3076923 (0.5491252) | 1.6923077 (0.8375789) | 1.5652174 (0.7277666)
  In the last 7 days, did you have any hair loss? | 1.0769231 (0.2717465) | 1.1153846 (0.4314555) | 1.6086957 (0.8913284)
  In the last 7 days, what was the severity of your problems with concentration at their worst? | 1.1923077 (0.4914656) | 1.5000000 (0.8602325) | 1.4782609 (0.7902569)
  In the past 7 days, how much did problems with concentration interfere with usual/daily activities? | 1.1538462 (0.543493) | 1.3076923 (0.6793662) | 1.3478261 (0.9820524)

ADVERSE EVENTS:
Time Frame: Adverse events were followed from start of treatment through 30 days after last dose of palbociclib.
Arm/Group | Palbociclib + Letrozole + Trastuzumab +/- Goserelin
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 2/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib + Letrozole + Trastuzumab +/- Goserelin (N=26)
Colonic obstruction (Gastrointestinal disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib + Letrozole + Trastuzumab +/- Goserelin (N=26)
Anemia (Blood and lymphatic system disorders) | 20
Intravenous antibiotics for positive blood cultures (Blood and lymphatic system disorders) | 1
Lymph node pain (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 2
Ventricular tachycardia (Cardiac disorders) | 1
Blurred vision (Eye disorders) | 3
Depth perception change (Eye disorders) | 1
Dry eye (Eye disorders) | 3
Stye - left eye (Eye disorders) | 1
Watering eyes (Eye disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 7
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 3
Hemorrhoids (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 8
Oral pain (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Stomach ache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Chills (General disorders) | 3
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 18
Fever (General disorders) | 1
Hypertension (General disorders) | 16
Left armpit pain (General disorders) | 1
Pain (General disorders) | 2
Right hip pain (General disorders) | 1
Right underarm edema (General disorders) | 1
Allergic reaction (Immune system disorders) | 1
Seasonal allergies (Immune system disorders) | 1
Bronchial infection (Infections and infestations) | 1
Cold sores (Infections and infestations) | 1
Papulopustular rash (Infections and infestations) | 1
Prophylactic herpes (Infections and infestations) | 1
Redness of nail bed - right (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Breast pain - surgery (Injury, poisoning and procedural complications) | 1
Pain related to surgery (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 6
Creatinine increased (Investigations) | 2
Ejection fraction decreased (Investigations) | 1
Electrocardiogram QT corrected (Investigations) | 1
Lymphocyte count decreased (Investigations) | 9
Neutrophil count decreased (Investigations) | 23
Platelet count decreased (Investigations) | 15
White blood cell decreased (Investigations) | 26
Anorexia (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Arthralgia - knees (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Concentration impairment (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 4
Headache (Nervous system disorders) | 11
Migraine (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy - fingers (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Bilateral breast pain (Reproductive system and breast disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Vaginal pruritus (Reproductive system and breast disorders) | 1
Cold/sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dry nose (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Runny nose (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Acne on nose (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Facial rash (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Itchy rash bilateral arms (Skin and subcutaneous tissue disorders) | 1
Mild rash face/chin (Skin and subcutaneous tissue disorders) | 1
Papular urticaria (Skin and subcutaneous tissue disorders) | 1
Peeling fingers (Skin and subcutaneous tissue disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculopapular (Skin and subcutaneous tissue disorders) | 3
Rash near port site (Skin and subcutaneous tissue disorders) | 1
Sensitive skin (Skin and subcutaneous tissue disorders) | 1
Skin pain (Skin and subcutaneous tissue disorders) | 1
Stye (Skin and subcutaneous tissue disorders) | 1
Hot flashes (Vascular disorders) | 5
Hypertension (Vascular disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT02907918/Prot_SAP_000.pdf